CLINICAL TRIAL: NCT01765491
Title: Comparison of Morning-only With Split-dose Polyethylene Glycol for Colonoscopy Preparation in Hospitalized Patients: A Randomized Controlled Non-Inferiority Study
Brief Title: Comparison of Two Methods of Bowel Preparation for Colonoscopy in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Bashar Attar MD, MD, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11-206
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: colonoscopy; bowel preparation; polyethylene glycol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morning-only polyethylene glycol (Experimental): One gallon of polyethylene glycol to be taken between 5am and 9am on the day of colonoscopy.
  Interventions: Other: Morning-only polyethylene glycol
- Split-dose polyethylene glycol (Active Comparator): Half gallon of polyethylene glycol to be taken between 7-9 pm on the day before colonoscopy and the remaining half between 7-9 am on the day of colonoscopy.
  Interventions: Other: Split-dose polyethylene glycol

INTERVENTIONS:
Other: Split-dose polyethylene glycol — Half gallon of polyethylene glycol to be taken between 7-9 pm on the day before colonoscopy and the remaining half between 7-9 am on the day of colonoscopy
  Arms: Split-dose polyethylene glycol
Other: Morning-only polyethylene glycol — One gallon of polyethylene glycol to be taken between 5am and 9am on the day of colonoscopy
  Arms: Morning-only polyethylene glycol

SUMMARY:
Morning-only colonoscopy preparation may improve efficiency by allowing same-day patient preparation and colonoscopy. The aim of the investigators study is to compare the efficacy and tolerability of morning-only Polyethylene Glycol (PEG) to split-dose preparation in hospitalized patients undergoing colonoscopy.

DETAILED DESCRIPTION:
This is a single-center, prospective, endoscopist-blinded study in which hospitalized patients scheduled to undergo diagnostic colonoscopy were randomly assigned to receive one gallon of PEG either the morning of colonoscopy or as a split-dose (evening-morning). The primary end point is efficacy of colonoscopy preparation measured by the Ottawa scale. The investigators pre-specified a non-inferiority margin of 1.5 for the difference in Ottawa scale between arms. Secondary end points are patient compliance and tolerance. N: 120 hospitalized patients scheduled for diagnostic colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo diagnostic colonoscopy during hospitalization

Exclusion Criteria:

* Critically ill/Intensive Care Unit patients
* Suspected bowel obstruction/perforation
* History of colon resection
* Patients with altered mental status/inability to provide informed consent
* Incarcerated patients
* Pregnant females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of colonoscopy preparation measured by the Ottawa scale | Day of procedure
  Colonoscopy was performed by gastroenterology fellows under the supervision of attending physicians and both were blinded to the type of preparation taken by the study patients. Bowel cleansing was evaluated by the Ottawa scale. Scoring of each part of the colon (right, middle and left) was done separately and the total amount of fluid was noted. The scores were then added to calculate the total score out of 14.

SECONDARY OUTCOMES:
Patient compliance | Day of procedure
  Before the patients were taken to the endoscopy suite, they completed a questionnaire, asking the amount of preparation that was taken to evaluate compliance.
Patient tolerance | Same day
  Before the patients were taken to the endoscopy suite, they completed a questionnaire to evaluate tolerance for taking the preparation. Patients were asked about side-effects like nausea, vomiting, abdominal pain and bloating.

CONTACTS AND LOCATIONS:
Overall Officials: Bashar Attar, MD, PhD, Study Director — Cook County Health & Hospitals System
Locations (1):
- John H Stroger Jr Hospital of Cook County, Chicago, Illinois, United States